CLINICAL TRIAL: NCT02450786
Title: Effect of Donepezil on Cognition in Parkinson's Disease With Mild Cognitive Impairment (PD-MCI)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-1089
Record Dates: First submitted 2015-05-14; First posted 2015-05-21 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Donepezil group (Experimental): Donepezil is started in 5mg for 8 weeks followed by dose escalation to 10mg and then maintained for 40 weeks. Participants who are not tolerable to dose of 10mg due to any issues of adverse effects would be maintained with donepezil 5mg exclusively in remained period.
  Interventions: Drug: Donepezil
- control group (No Intervention): No administration of any therapeutic medications for dementia including cholinesterase inhibitor or NMDA receptor blocking agents. Standard treatment protocol of Parkinson's disease with mild cognitive impairment would be fulfilled including dopaminergic or nondopaminergic medications as well as nootropic drugs.

INTERVENTIONS:
Drug: Donepezil — Donepezil is started in patients with Parkinson's disease mild cognitive impairment with 5mg for 8 weeks followed by dose up to 10mg and then maintained for 40 weeks. Participants who are not tolerable to dose of 10mg due to any issues of adverse effects would be maintained with donepezil 5mg exclusively in remained period.
  Arms: Donepezil group

SUMMARY:
There have been growing interest in identifying Parkinson's disease (PD) patients with mild cognitive impairment (MCI) which is susceptible to progress to PD dementia(PDD). PD-MCI is known to significantly correlates with low cerebrospinal beta-amyloid 1-42 and 1-40 levels, in which suggest the existence of something common with Alzheimer's dementia. PDD have showed more cholinergic deficits than Alzheimer's dementia and responds to donepezil. The investigators assume that PD-MCI patients also have cholinergic deficits. Donepezil improves cognition, and seems to be well tolerated and not to worsen parkinsonism in patients with cognitive impairment. Donepezil produced similar improvements in cognition and behaviour in DLB and PDD. This supports the hypothesis that the two disorders are closely related clinically and neurobiologically. Larger scale, placebo controlled clinical trials are needed to provide an evidence base to guide the clinical use of cholinesterase inhibitors in Lewy body disease.

It is believed that earlier intervention, later appearance of dementia should be needed to lower the socioeconomic costs and to improve the quality of life on patients and caregivers. The investigators anticipate that donepezil may delay the development of dementia in patients with PD-MCI.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 40 years old
* Clinical diagnosis of PD established by Queen Square Brain Bank Criteria
* Stable dose of levodopa at least 3 months before the study enrollment
* Diagnosis of MCI in PD according to the Movement Disorder Society (MDS) task force guideline

Exclusion Criteria:

* Diagnosis of Dementia
* Hypersensitivity to piperidine derivatives
* Concomitant anticholinergics and cholinergic agents
* Severe cardiac arrhythmia: Sick sinus syndrome, complete AV block, Uncontrolled arrhythmia, history of ventricular fibrillation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Rate of cognitive decline | at 48wks
  Korean Version of Mini-Mental State Exam

SECONDARY OUTCOMES:
changes of cognitive decline | baseline, 24 wks, 48 wks, 72 wks
changes of Parkinson's disease motor scale | baseline, 24 wks, 48 wks, 72wks
  UPDRS part I-IV
Brain structure (cortical thickness and subcortical volume/shape) and Default mode network | 48wks
  Conventional and functional brian MRI
brain functional connectivity | 48wks
  digital electroencephalography
Comprehensive neuropsychological test | 48wks
  Seoul Neuropsychological Screening Battery (SNSB)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea